CLINICAL TRIAL: NCT02205294
Title: The Effect of Osteopathic Treatment in Acute Proximal Leg Deep Vein Thrombosis (DVT) to Reduce Pain and Swelling
Brief Title: Osteopathic Treatment and Deep Vein Thrombosis (DVT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REB ROMEO # 1017573
Record Dates: First submitted 2014-07-29; First posted 2014-07-31 (Estimated); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Deep Vein Thrombosis (DVT)
Keywords: Osteopathic treatment; Deep Vein Thrombosis; Proximal Leg DVT
MeSH Terms: conditions — Venous Thrombosis | interventions — Manipulation, Osteopathic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Assessment Only (No Intervention): Subjects will have an osteopathic assessment to determine areas of tension in specific areas of the body. These areas include: the thoracic diaphragm, the heart and pericardium, the iliac fascia, the femoral sheath, the sartorius muscle, the pelvic diaphragm and the interosseous membrane (IM) of the lower extremity
- Assessment and Treatment (Active Comparator): Subjects will have an osteopathic assessment to determine areas of tension in specific areas of the body. These areas of tension will receive osteopathic treatment, using myofascial release techniques. These areas include: the thoracic diaphragm, the heart and pericardium, the iliac fascia, the femoral sheath, the sartorius muscle, the pelvic diaphragm and the interosseous membrane (IM) of the lower extremity
  Interventions: Other: Osteopathic Treatment

INTERVENTIONS:
Other: Osteopathic Treatment — The osteopathic treatment will be a gentle hands treatment using myofascial release techniques.
  Arms: Assessment and Treatment

SUMMARY:
Osteopathic treatment will provide:

1. A significant reduction of pain and swelling of the affected DVT leg
2. An increase in the quality of life (QOL) for individuals with DVT of the leg
3. Improved signs and symptoms of the post thrombotic syndrome of the affected DVT leg

DETAILED DESCRIPTION:
Thousands of individuals are affected by deep vein thrombosis (DVT) every year. Medical treatment is aimed at preventing extension and recurrence of the blood clot (DVT) through the use of anticoagulation medication. Compression stockings may be added for reduction of pain and swelling, but this therapy remains controversial amongst physicians. To date, there is limited manual therapies available for individuals affected with DVT. Regular medical treatment, anticoagulation medication, along with osteopathic treatment may offer these individuals improved control of the symptoms associated with DVT. In the long term osteopathic treatment may provide an increase in the quality of life (QOL) and improve the signs and symptoms associated with the post-thrombotic syndrome (PTS), which can be burdensome for both the individual and the health care system. Offering an effective add on treatment could provide individuals and the medical system with an additional means of treatment for the symptoms of DVT and also for the prevention of development of PTS.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* first episode of symptomatic objectively confirmed proximal leg DVT without pulmonary embolism
* 1 month of appropriate anticoagulation treatment
* therapeutic level of anticoagulation (ie: Warfarin, INR- 2.0-3.0)

Exclusion Criteria:

* > 1 month + 7 days of anticoagulation
* history of previously confirmed proximal or distal leg DVT
* medically unstable individuals requiring hospitalization
* history of peripheral vascular disease (PVD)
* injury of affected leg (trauma within the last 6 months or leg currently casted)
* history of previous stroke
* uncontrolled hypertension
* renal failure requiring hemodialysis or peritoneal dialysis
* diagnosis of cancer in the last five years or currently receiving treatment for cancer
* open heart or vascular surgery in the last year
* any neurological condition (ie: MS, ALS, Parkinsons, etc)
* currently pregnant
* geographic inaccessibility
* unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-11-06 (Actual); Primary Completion 2019-04-04 (Actual); Study Completion 2019-04-04 (Actual)

PRIMARY OUTCOMES:
Swelling | 1 month pre and post testing and 2 months
  Swelling will be measured using a tension-controlled tape measure at the initial study visit, one month after diagnosis of the subject's DVT and then again at 2 months after diagnosis.

SECONDARY OUTCOMES:
Leg Pain | 1 month pre and post testing and 2 months
  Leg Pain will be measured using the visual analogue scale (VAS), at the initial study visit(1 month after diagnosis of the DVT) pre and post assessment or assessment plus treatment. Pain will be evaluated again at the 2 month visit post answering questionnaires and lying supine for 10 minutes.

OTHER OUTCOMES:
Quality of LIfe (QOL) | 1 month and 2 months
  Veines QOL/Sym Questionnaire will be completed by all participants at both study visits to determine if there have been any changes.
Assessment for Post Thrombotic Syndrome (PTS) | 1 month and 2 months
  The Villalta scale will be used to assess subjects for signs and symptoms of the post-thrombotic syndrome at both study visits.

CONTACTS AND LOCATIONS:
Overall Officials: Darlene D MacLeod, BscN DOMP, Principal Investigator — Nova Scotia Health Authority
Locations (1):
- QEll Health Sciences Centre, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: Undecided
Pending numbers recruited